CLINICAL TRIAL: NCT01169298
Title: A Phase I, Multicenter, Open-label, Dose-escalation Study to Assess the Safety of Lenalidomide in Patients With Advanced Adult T-cell Leukemia-lymphoma and Peripheral T-cell Lymphoma
Brief Title: A Phase I, Multicenter, Open-label, Dose-escalation Study to Assess the Safety of Lenalidomide in Patients With Advanced Adult T-cell Leukemia-lymphoma and Peripheral T-cell Lymphomaperipheral T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-ATLL-001
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Adult T-cell Leukemia-Lymphoma; Peripheral T-cell Lymphoma
Keywords: Adult T-cell Leukemia-Lymphoma; Peripheral T-cell Lymphoma; PTCL; HTLV-1
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Lymphoma, T-Cell, Peripheral | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide: 25mg daily on day1-21 of each 28days cycle (1st cohort), 25 mg daily of each 28 days (2nd cohort) or 35 mg daily of each 28 days (3rd cohort)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide: 25mg daily on day 1-21 of each 28days cycle (1st cohort), 25 mg daily of each 28 days (2nd cohort, or 35 mg daily of each 28 days (3rd cohort)

SUMMARY:
To determine the maximum tolerated dose of lenalidomide in patients with adult T-cell leukemia-lymphoma (ATL) and peripheral T-cell lymphoma (PTCL) who have previously received therapy for ATL and PTCL

ELIGIBILITY:
Inclusion Criteria:

1. Subject must understand and voluntarily sign the written informed consent;
2. Aged 20 years or older;
3. Subject have a documented diagnosis of either:

   * Acute-, lymphoma-, or unfavorable chronic-type ATL or
   * Peripheral T-cell Lymphomaperipheral (PTCL)
4. Subject have received ≥1 prior anti-cancer therapy, have achieved stable disease (SD) or better on their immediately prior therapy and have relapsed or progressed at the time of obtaining signed informed consent;
5. Subject have an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 2 at enrollment;

Exclusion Criteria:

1. Natural Killer cell lymphoma (NK-cell lymphoma);
2. T-cell leukemia;
3. Cutaneous T-cell lymphoma (CTCL) including;

   * Mycosis fungoides
   * Sezary syndrome
   * CD30-positive lympho-proliferative disorders
   * Cutaneous gamma/delta T-cell lymphoma
4. Subject have a history of central nervous system (CNS) involvement or present with CNS symptoms, and are diagnosed with CNS lymphoma by cerebrospinal fluid (CSF) cytology examination, head CT scan or brain MRI during the screening;
5. Are pregnant or lactating;
6. Subject have uncontrolled inter-current illness including:

   * Uncontrolled diabetes mellitus
   * Chronic congestive heart failure (NYHA Class III or IV)
   * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction (within 6 months before starting the study drug)
   * Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia
   * Other uncontrolled diseases
7. Exhibit grade 4 neurological disorders;
8. Subject have a history or complication of deep vein thrombosis or pulmonary embolism within 6 months before the start of study treatment;
9. Develop active tuberculous disease, herpes simplex, systemic mycosis, or other active infections requiring systemic administration of antibiotics, antiviral agents, or antifungal drugs;
10. Are tested positive for HBs antigen, anti-HCV antibody, or anti-HIV antibody;
11. Subjects have a history or complication for which the investigator or subinvestigator deems them inappropriate for this study, or have serious diseases or mental illness that is likely to be aggravated by participation in this study;
12. Subjects have a history of allogeneic stem cell transplantation;
13. Subjects have received autologous stem cell transplantation within 12 weeks (84 days) of the start of study treatment;
14. Have previously used lenalidomide;
15. Have a history of desquamating (bullous) rash while taking thalidomide;
16. Have received any investigational drugs (unapproved drugs in Japan) within 4 weeks (28 days) of the start of study medication;
17. Have received chemotherapeutic agents or immunomodulators for the treatment of ATL or PTCL within 4 weeks (28 days) of the start of study treatment;
18. Have received radiotherapy within 4 weeks (28 days) of the start of study treatment;
19. Have a history or complication of another malignant tumor than ATL or PTCL (excluding malignant tumors below), unless the patients have been free of the disease for 5 years or longer;

    * Cutaneous basal cell carcinoma or squamous cell carcinoma
    * Cervical carcinoma in situ
    * An incidental histological finding of prostate carcinoma (TNM stage T1a or T1b)
20. Have had any of the following abnormal measurements at screening performed within 1 week (7 days) prior to the enrollment;

    * Neutrophil count: < 1,200/µL (1.2 x 109/L)
    * Platelet count: < 75,000/µL (75 x 109/L)
    * Serum aspartate aminotransferase/ Serum glutamic oxaloacetic transaminase (AST/SGOT) or Alanine transaminase/Serum Glutamic Pyruvate Transaminase (ALT/SGPT): > 3 times the Upper Limit of Normal (ULN)
    * Bilirubin level: > 1.5 times of the ULN
    * Creatinine clearance: < 60 mL/min

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-20 (Actual)

PRIMARY OUTCOMES:
The safety of lenalidomide evaluated based on the severity of adverse events and their causality | Up to 2.5 years
  The safety of lenalidomide evaluated based on the severity of adverse events and their causality

SECONDARY OUTCOMES:
Response | Up to 2.5 years
  The response of ATL patient to lenalidomide will be evaluated according to the criteria proposed by the International Consensus Meeting.
  The response of PTCL will be assessed by the Japan Clinical Oncology Group (JCOG) response criteria that have been established by the Lymphoma Study Group of the JCOG based on criteria of Cheson et al.in the Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas
PK-Time to Maximum Plasma Concentration (Tmax) | Day 8 of Cycle 1
  PK-Time to Maximum Plasma Concentration (Tmax)
PK-Apparent Total Body Clearance (CL/F) | Day 8 of Cycle 1
  PK-Apparent Total Body Clearance (CL/F)
PK-Apparent Volume of Distribution (Vz/F) | Day 8 of Cycle 1
  PK-Apparent Volume of Distribution (Vz/F)
PK-Terminal half-life (T1/2) | Day 8 of Cycle 1
  PK-Terminal half-life (T1/2)
PK-Area under the Plasma concentration time curve (AUC) | Day 8 of Cycle 1
  PK-Area under the Plasma concentration time curve (AUC)
Accumulation ratio (Cmax) | Day 8 of Cycle 1
  Accumulation ratio (Cmax)
Accumulation ratio (AUCτ) | Day 8 of Cycle 1
  Accumulation ratio (AUCτ)
PK-Maximum Concentration in Plasma (Cmax) | Day 8 of cycle 1
  PK-Maximum Concentration in Plasma (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroya Asou, MD, Study Director — Celgene KK
Locations (6):
- Japan (6):
  - National Kyusyu Cancer Center, Fukuoka
  - Imamura Bun-in Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - Nagoya Daini Red Cross Hospital, Nagoya
  - National Cancer Center Hospital, Tokyo

REFERENCES:
- [Background] Ogura M, Imaizumi Y, Uike N, Asou N, Utsunomiya A, Uchida T, Aoki T, Tsukasaki K, Taguchi J, Choi I, Maruyama D, Nosaka K, Chen N, Midorikawa S, Ohtsu T, Tobinai K. Lenalidomide in relapsed adult T-cell leukaemia-lymphoma or peripheral T-cell lymphoma (ATLL-001): a phase 1, multicentre, dose-escalation study. Lancet Haematol. 2016 Mar;3(3):e107-18. doi: 10.1016/S2352-3026(15)00284-7. Epub 2016 Feb 12. PMID 26947199